CLINICAL TRIAL: NCT00697346
Title: An Open-label, Phase 1 Study of MLN8237, a Novel Aurora A Kinase Inhibitor, in Patients With Advanced Hematological Malignancies
Brief Title: Study of MLN8237 in Participants With Advanced Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C14003; U1111-1187-1184 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: B-cell Follicular Lymphoma; B-cell Marginal Zone Lymphoma; Diffuse Large B-cell Lymphoma; B-cell Mantle Cell Lymphoma; B-cell Small Lymphocytic Lymphoma; B-Cell Chronic Lymphocytic Leukemia; Multiple Myeloma; Waldenstrom's Macroglobulinemia; Noncutaneous Peripheral T-cell Lymphoma Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Enteropathy Associated T-cell Lymphoma; NK Lymphoma
Keywords: Drug therapy
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Enteropathy-Associated T-Cell Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: PIC Dose Escalation (Experimental): Alisertib 25 or 35 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 21 days followed by a 7-day recovery period in 28-day cycles or alisertib 35, 45, 65 or 90 mg PIC, orally, (QD for 14 days followed by a 14-day recovery period in 28-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 14 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose), followed by their respective dosage assignment.
  Interventions: Drug: Alisertib
- Part 1: ECT Dose Escalation (Experimental): Alisertib 40 mg, Enteric-coated Tablet (ECT) formulation, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, or alisertib 30, 40 or 50 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 15 cycles).
  Interventions: Drug: Alisertib
- Part 2: PTCL (Experimental): Participants with peripheral T-cell lymphoma (PTCL) received alisertib 50 mg ECT, orally, BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib (MLN8237) PIC or ECT
  Other Names: MLN8237

SUMMARY:
This is an open-label, multicenter, phase 1 study of MLN8237 in participants with advanced hematological malignancies for whom there are limited standard treatment options.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib. Alisertib is being tested to treat people who have advanced hematological malignancies. This study determined the dose-limiting toxicity, maximum tolerated dose, safety and pharmacokinetics (how the drug moves through the body) for alisertib when given once or twice a day for 7 to 21 days.

This open label study enrolled 58 patients. Participants were enrolled in one of 3 treatment groups:

* Part 1: Powder-in-Capsule (PIC) Dose Escalation (alisertib 25 mg PIC, orally twice daily [BID] on Day 1 [loading dose] and then alisertib 25 or 35 mg PIC once daily [QD] for 21 days (D), or alisertib 35, 45, 65 or 90 mg PIC, orally, QD for 14D) in 28-day cycles
* Part 1: Enteric-coated Tablet (ECT) Dose Escalation (alisertib 40 mg, ECT, orally, QD for 14D or alisertib 30, 40 or 50 mg, orally, BID for 7D) in 28-day cycles
* Part 2: Participants with Peripheral T-cell Lymphoma (PTCL) (alisertib 50 mg ECT, orally, BID for 7D) in 21-day cycles

All participants received treatment for 12 months or until their disease progressed or they experienced unacceptable alisertib-related toxicity. This multi-center trial was conducted in the United States. The overall time to participate in this study was 422 days. Participants made multiple visits to the clinic, including a final visit 30 days after receiving their last dose of alisertib for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory disease and a histologically or cytologically confirmed hematological malignancy of the following type for which standard curative treatment does not exist or is no longer effective:

  * B-cell Follicular lymphoma
  * B-cell Marginal zone lymphoma
  * Diffuse large B-cell lymphoma
  * B-cell Mantle cell lymphoma
  * B-cell Small lymphocytic lymphoma (SLL)
  * B-Cell Chronic lymphocytic leukemia (B-CLL)
  * Multiple myeloma
  * Waldenstrom's macroglobulinemia
  * Noncutaneous peripheral T-cell lymphoma not otherwise specified (PTCL-NOS)
  * Angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma, enteropathy associated T-cell lymphoma (EATCL), NK lymphoma (NKL)
* Participants with diffuse large B-cell lymphoma must have failed, be ineligible for, or have refused an autologous stem cell transplant. There is no restriction regarding the maximum number of prior regimens.
* Aged 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Radiographically or clinically evaluable disease for Part 1 of this study and measurable disease for Part 2 of this study
* Suitable venous access for the conduct of blood sampling for MLN8237 pharmacokinetics (PK)
* Recovered from the reversible effects of prior antineoplastic treatment (with the exception of alopecia and Grade 1 neuropathy)

Exclusion Criteria:

* Pregnant or lactating
* Treatment with clinically significant enzyme inducers within 14 days prior to the first dose of MLN8237 as specified in the protocol
* Prior allogeneic bone marrow (or other organ) transplantation
* Newly diagnosed or uncontrolled cancer-related central nervous system (CNS) disease
* Systemic antineoplastic treatment within 21 days preceding the first dose of study treatment. Exceptions requiring a 42-day recovery period from last treatment include: Nitrosoureas, mitomycin C or Rituximab, alemtuzumab (Campath®), or other unconjugated therapeutic antibody (21 days if clear evidence of progressive disease)
* Treatment with radioimmunoconjugates or toxin immunoconjugates such as ibritumomab tiuxetan (Zevalin™), or tositumomab (Bexxar®) within 56 days preceding the first dose of study treatment
* Antineoplastic treatment with glucocorticoids within 21 days preceding the first dose of study treatment
* Radiotherapy involving <25% of the hematopoietically active bone marrow within 21 days preceding first dose of study treatment
* Radiotherapy involving ≥25% of the hematopoietically active bone marrow within 42 days preceding first dose of study treatment
* Inability to swallow capsules or known gastrointestinal (GI) disease or GI procedures that could interfere with the oral absorption or tolerance of MLN8237. Examples include, but are not limited to, partial gastrectomy, history of small intestine surgery, and celiac disease.
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection. Testing is not required in the absence of clinical findings or suspicion.
* Participants who fail to meet laboratory values as specified in the protocol during the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - Scottsdale, Arizona
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Buffalo, New York
  - Chapel Hill, North Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Kelly KR, Shea TC, Goy A, Berdeja JG, Reeder CB, McDonagh KT, Zhou X, Danaee H, Liu H, Ecsedy JA, Niu H, Benaim E, Iyer SP. Phase I study of MLN8237--investigational Aurora A kinase inhibitor--in relapsed/refractory multiple myeloma, non-Hodgkin lymphoma and chronic lymphocytic leukemia. Invest New Drugs. 2014 Jun;32(3):489-99. doi: 10.1007/s10637-013-0050-9. Epub 2013 Dec 20. PMID 24352795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 11 July 2008 to19 October 2016.
Pre-assignment Details: Participants with a diagnosis of advanced hematological malignancies were enrolled 1 of 3 treatment groups, Part 1:alisertib powder-in capsule (PIC) 25 to 90 mg dose escalation cohort, Part 1: alisertib 30 to 50 mg enteric-coated tablet (ECT) dose escalation cohort, or Part 2: alisertib ECT 50 mg participants with peripheral T-cell lymphoma (PTCL).
Groups:
- Part 1: PIC Dose Escalation: Alisertib 25 or 35 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 21 days followed by a 7-day recovery period in 28-day cycles or alisertib 35, 45, 65 or 90 mg PIC, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 14 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose), followed by their respective dosage assignment.
Period: Overall Study
Arm/Group | Part 1: PIC Dose Escalation | Part 1: ECT Dose Escalation | Part 2: PTCL
Started | 28 | 28 | 2
Completed | 0 (Completed = participants who completed study treatment.) | 2 (2 participants were ongoing as of primary completion date 27 Dec 2011 and have now completed.) | 1 (1 participant was ongoing as of primary completion date 27 Dec 2011 and has now completed.)
Not Completed | 28 | 26 | 1
Not completed — Adverse Event | 4 | 5 | 0
Not completed — Progressive Disease | 19 | 18 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Reason not Specified | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population is defined as all participants who received any amount of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: PIC Dose Escalation | Part 1: ECT Dose Escalation | Part 2: PTCL | Total
Number analyzed (Participants) | 28 | 28 | 2 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.91) | 59.5 (14.22) | 63.0 (24.04) | 60.5 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 2 | 31
  Male | 14 | 13 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 0 | 16
  Not Hispanic or Latino | 19 | 20 | 2 | 41
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 26 | 2 | 52
  Black or African American | 3 | 1 | 0 | 4
  Asian | 0 | 1 | 0 | 1
  Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 2 | 58
Height [Mean (Standard Deviation); unit: cm] — Population: Here number analyzed is the number of participants who were evaluated for height at baseline.
  cm
    number analyzed (Participants) | 28 | 26 | 2 | 56
    (all) | 165.9 (11.25) | 164.6 (10.95) | 160.6 (6.43) | 165.1 (10.89)
Weight [Mean (Standard Deviation); unit: kg] | 81.40 (20.031) | 77.62 (19.747) | 97.65 (43.911) | 80.13 (20.573)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body Surface Area =square root [height (cm) * weight (kg) / 3600]. Population: Here number analyzed is the number of participants who were evaluated for body surface area at baseline.
  m^2
    number analyzed (Participants) | 28 | 26 | 2 | 56
    (all) | 1.93 (0.282) | 1.88 (0.289) | 2.05 (0.434) | 1.91 (0.286)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and was defined as any of the following events related to therapy with alisertib:1. Grade 4 neutropenia lasting ≥7 consecutive days, 2. Grade 4 neutropenia with fever and/or infection 3. Platelet count <25,000/mm^3 4. Grade 3 or greater nausea and/or emesis despite use of optimal antiemetic prophylaxis 5. Grade 3 or greater diarrhea despite maximal supportive therapy with loperamide 6. Any other Grade 3 or greater nonhematologic toxicity, with the following exceptions: Grade 3 arthralgia/myalgias, Any grade of alopecia, Brief (<1 week) Grade 3 fatigue 7. Treatment delay of >21 days due to failure of adequate hematologic or non-hematologic recovery from previous cycle of treatment 8. Other alisertib related non-hematologic toxicities ≥Grade 2 that, in the opinion of the investigator required a dose reduction or discontinuation of therapy with alisertib.
Time Frame: From first dose of study drug to 30 days after the last dose (up to 422 days)
Population: DLT evaluable population included all participants who received at least 75% of their planned alisertib doses for their first cycle of treatment (unless interrupted by DLT) and had sufficient follow up data to allow the investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Groups:
- Alisertib 25mg PIC QD 21D: Alisertib 25 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 21 days (D) followed by a 7-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 35 mg PIC QD 21D: Alisertib 35 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 21 days followed by a 7-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 35 mg PIC QD 14D: Alisertib 35 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 14 days followed by a 14-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 45 mg PIC QD 14D: Alisertib 45 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 14 days followed by a 14-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity to (up 4 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 65 mg PIC QD 14D: Alisertib 65 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 14 days followed by a 14-day recovery period in 28-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 90 mg PIC QD 14D: Alisertib 90 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 14 days followed by a 14-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity (up to 5 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 40 mg ECT QD 14D: Alisertib 40 mg, Enteric-coated Tablet (ECT) formulation, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles until disease progression or unacceptable alisertib-related toxicity (up to 3 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 30 mg ECT BID 7D: Alisertib 30 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 40 mg ECT BID 7D: alisertib 40 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
- Alisertib 50 mg ECT BID 7D: Alisertib 50 mg ECT, orally BID for 7 Ddays followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D | Alisertib 90 mg PIC QD 14D | Alisertib 40 mg ECT QD 14D | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 6 | 4 | 3 | 6 | 6 | 2 | 4 | 3 | 7 | 9
participants | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Alisertib
Description: MTD was defined as the highest dose at which DLT occurred in 0/3 or 1/6 participants.
Time Frame: From first dose of study drug to 30 days after the last dose (up to 422 days)
Population: as for outcome 1
Measure: Number; unit: mg BID for 7 days
Groups:
- Alisertib: Alisertib 25 or 35 mg, PIC formulation, orally, once daily (QD) for 21 days followed by a 7-day recovery period in 28-day cycles or alisertib 35, 45, 65 or 90 mg PIC, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 14 cycles) followed by alisertib 50 mg ECT, orally, BID for 7 days followed by a 14-day recovery period in 21-day cycles or alisertib 40 mg, ECT formulation, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, or alisertib 30, 40 or 50 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity alisertib 50 mg ECT, orally, BID for 7 days followed by a 14-day recovery period in 21-day cycles (up to 14 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
Arm/Group | Alisertib
Number analyzed (Participants) | 58
mg BID for 7 days | 50

3. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: Pharmacokinetic (PK) evaluable population included all participants for whom there were sufficient dosing and alisertib concentration time data to permit non-compartmental PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 4
nM | 833.2 (49.5) | 1078.3 (26.4)

4. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple timepoints (up to 6 hours) postdose
Population: PK evaluable population included all participants for whom there were sufficient dosing and alisertib concentration time data to permit non-compartmental PK analysis. Here number of participants analyzed were participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
nM | 1337.6 (57.8) | 1451.9 (26.2)

5. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 4
hours (h) | 2.0 [2.0 to 3.3] | 2.0 [1.1 to 5.2]

6. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple timepoints (up to 6 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
h | 2.0 [1.0 to 5.0] | 2.0 [2.0 to 2.0]

7. Primary Outcome: AUCt: Area Under the Concentration Time Curve From Time 0 to Time t for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple time points (up to 6 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
nM*h | 14846 (69.7) | 16528 (35.6)

8. Primary Outcome: Terminal Half-Life (t1/2) for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple time points (up to 6 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 5 | 3
h | 20.5 (7.3) | 19.5 (6.0)

9. Primary Outcome: Accumulation Ratio (Rac) for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple time points (up to 6 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
ratio | 1.9 (1.1) | 1.5 (0.5)

10. Primary Outcome: Peak/Trough Ratio for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple timepoints (up to 6 hours) postdose
Population: PK evaluable population included all participants for whom there were sufficient dosing and alisertib concentration time data to permit non-compartmental PK analysis, with data available at the given time point. Here number of participants analyzed were participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
ratio | 6.0 (4.4) | 4.3 (1.5)

11. Primary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Pill in Capsule (PIC) With Once Daily for 21 Days (QD21D) Dosing at Day 21
Time Frame: Cycle 1 Day 21 predose and at multiple timepoints (up to 6 hours) postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Alisertib 25mg PIC QD 21D | Alisertib 35 mg PIC QD 21D
Number analyzed (Participants) | 6 | 3
L/h | 3.2 (113) | 4.1 (45)

12. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: PK evaluable population included all participants for whom there were sufficient dosing and alisertib concentration time data to permit non-compartmental PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D | Alisertib 90 mg PIC QD 14D
Number analyzed (Participants) | 3 | 6 | 7 | 2
nM | 726.5 (34.8) | 1637.0 (58.0) | 1773.4 (44.3) | 2497.4 (24.3)

13. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
nM | 2193.5 (NA) — Geometric Coefficient of Variation was not calculated for 2 participants. | 1634.4 (52.5) | 2300.2 (40.3)

14. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 12
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D | Alisertib 90 mg PIC QD 14D
Number analyzed (Participants) | 3 | 6 | 7 | 2
h | 2.0 (34.8) [1.9 to 4.0] | 3.0 (58.0) [1.1 to 4.0] | 2.0 (44.3) [1.9 to 6.0] | 2.9 (24.3) [1.5 to 4.3]

15. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
h | 3.4 (NA) [0.8 to 6.1] | 2.0 (52.5) [2.0 to 4.0] | 2.0 (40.3) [1.5 to 2.1]

16. Primary Outcome: AUCt: Area Under the Concentration Time Curve From Time 0 to Time t for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
nM*h | 23444 (NA) [1.9 to 4.0] — Geometric Coefficient of Variation was not calculated for 2 participants. | 19671 (64.8) [1.1 to 4.0] | 28864 (39.9) [1.9 to 6.0]

17. Primary Outcome: Accumulation Ratio (Rac) for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
ratio | 2.4 (0.00) [1.9 to 4.0] | 1.5 (0.5) [1.1 to 4.0] | 1.9 (1.6) [1.9 to 6.0]

18. Primary Outcome: Peak/Trough Ratio for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
ratio | 4.1 (NA) [1.9 to 4.0] — Standard deviation was not calculated for 2 participants. | 5.4 (1.9) [1.1 to 4.0] | 4.4 (0.8) [1.9 to 6.0]

19. Primary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Pill in Capsule (PIC) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Alisertib 35 mg PIC QD 14D | Alisertib 45 mg PIC QD 14D | Alisertib 65 mg PIC QD 14D
Number analyzed (Participants) | 2 | 5 | 6
L/h | 2.9 (NA) [1.9 to 4.0] — Geometric Coefficient of Variation was not calculated for 2 participants. | 4.3 (44) [1.1 to 4.0] | 4.3 (53) [1.9 to 6.0]

20. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 6
nM | 1227 (41.3)

21. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: PK evaluable population included all participants for whom there were sufficient dosing and alisertib concentration time data to permit non-compartmental PK analysis. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 2
nM | 1608 (NA) — Geometric Coefficient of Variation was not calculated for 2 participants.

22. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 24 hours) postdose
Population: as for outcome 12
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 6
h | 3.9 (NA) [2.0 to 6.1]

23. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 21
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 2
h | 5.0 (NA) [4.0 to 6.0]

24. Primary Outcome: AUCt: Area Under the Concentration Time Curve From Time 0 to Time t for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 5
nM*h | 14306 (20.3) [2.0 to 6.1]

25. Primary Outcome: Terminal Half Life for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 1
h | 11.7 (NA) [2.0 to 6.1] — Standard deviation is not estimable for 1 participant.

26. Primary Outcome: Peak/Trough Ratio for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 1
ratio | 2.1 (NA) [2.0 to 6.1] — Standard deviation is not estimable for 1 participant.

27. Primary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Enteric Coated Tablet (ECT) With Once Daily for 14 Days (QD14D) Dosing at Day 14
Time Frame: Cycle 1 Day 14 predose and at multiple timepoints (up to 8 hours) postdose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Alisertib 40 mg ECT QD 14D
Number analyzed (Participants) | 1
L/h | 2.5 (NA) [2.0 to 6.1] — Standard deviation is not estimable for 1 participant.

28. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Alisertib 50 mg ECT BID 7D: Alisertib 50 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 6 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose).
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 9 | 10
nM | 886 (39.7) | 1114 (37.1) | 1531 (58.4)

29. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 8 | 7
nM | 2025 (29.6) | 2586 (35.7) | 2058 (44.6)

30. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 1
Time Frame: Cycle 1 Day 1 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 9 | 10
h | 2.0 (39.7) [2.0 to 2.0] | 2.2 (37.1) [2.0 to 6.0] | 2.0 (58.4) [2.0 to 8.0]

31. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 8 | 7
h | 2.0 (39.7) [2.0 to 2.0] | 2.2 (37.1) [1.0 to 3.6] | 2.0 (58.4) [1.3 to 6.0]

32. Primary Outcome: AUCt: Area Under the Concentration Time Curve From Time 0 to Time t for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 1
Time Frame: Cycle 1 Days 1 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 9 | 9
nM*hr | 5518 (18.3) | 7095 (42.5) | 9732 (48.5)

33. Primary Outcome: AUCt: Area Under the Concentration Time Curve From Time 0 to Time t for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 8 | 7
nM*hr | 16024 (20.3) | 18624 (27.3) | 17914 (48.6)

34. Primary Outcome: Terminal Half-Life (t1/2) for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 1 | 4 | 5
h | 13.3 (NA) — Standard deviation was not calculated for 2 participants. | 19.9 (10.7) | 18.4 (13.9)

35. Primary Outcome: Accumulation Ratio (Rac) for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 7 | 6
ratio | 2.9 (0.5) | 2.8 (1.0) | 2.3 (0.9)

36. Primary Outcome: Peak/Trough Ratio for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 7 | 7
ratio | 2.5 (0.6) | 2.4 (0.5) | 2.5 (2.2)

37. Primary Outcome: CLss/F: Apparent Oral Clearance at Steady State for Alisertib as Enteric Coated Tablet (ECT) With Twice Daily for 7 Days (BID7D) Dosing at Day 7
Time Frame: Cycle 1 Day 7 predose and at multiple timepoints (up to 12 hours) postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Alisertib 30 mg ECT BID 7D | Alisertib 40 mg ECT BID 7D | Alisertib 50 mg ECT BID 7D
Number analyzed (Participants) | 3 | 7 | 7
L/h | 3.7 (0.7) | 4.4 (1.9) | 6.7 (5.6)

38. Secondary Outcome: Best Overall Response Rate Based on Investigator's Assessment
Description: Best overall response rate is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the Investigator using International Working Group (IWG) Criteria. CR is defined as the disappearance of all evidence of disease and the definition for PR includes at least a 50% decrease in sum of the product of the diameters and no new lesions.
Time Frame: Baseline and every 2 cycles up to Month 12 until disease progression, 30 days after end of treatment (up to 422 days)
Population: The response-evaluable population is defined as all participants who received at least 1 dose of alisertib and have measurable disease at baseline and have at least 1 post baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: PIC Dose Escalation | Part 1: ECT Dose Escalation | Part 2: PTCL
Number analyzed (Participants) | 23 | 23 | 1
percentage of participants | 13 | 9 | 100

39. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a response (either CR or PR) to the date of first documentation of progressive disease (PD) according to International Working Group (IWG) criteria. CR is defined as the disappearance of all evidence of disease and the definition for PR includes at least a 50% decrease in sum of the product of the diameters and no new lesions. PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Baseline and every 2 cycles up to Month 12 until disease progression, 30 days after end of treatment (up to 422 days)
Population: Participants from the Response-Evaluable Population who had a response of CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Part 1: PIC Dose Escalation | Part 1: ECT Dose Escalation | Part 2: PTCL
Number analyzed (Participants) | 3 | 2 | 1
months | 0.03 [0.03 to 3.65] | 2.07 [0.03 to 4.18] | 0.03 [0.03 to 0.03]

40. Secondary Outcome: Number of Participants With Polymorphisms in Gene Encoding Enzyme UGT1A1
Description: One peripheral blood sample (approximately 4 mL) was to be obtained on Day 1 of Cycle 1 prior to the first dose of alisertib to genotype participants for polymorphisms in UGT1A1 because UGT1A1 is one of the enzymes responsible for glucuronidation of alisertib, which is expected to contribute to the clearance of alisertib.
  wt=wild type. *28=polymorphism in the promoter region of a UGT1A1 allele resulting in reduced UGT1A1 expression. Not determined = blood sample was not evaluable.
Time Frame: Cycle 1 Day 1 predose
Population: Safety population included all participants who received any amount of study drug. Data is presented for one arm because the data was collected prior to the participant receiving their assigned treatment.
Measure: Number; unit: participants
Arm/Group | Alisertib
Number analyzed (Participants) | 58
participants
  wt/wt | 23
  wt/*28 | 23
  *28/*28 | 8
  other/other | 1
  Not Determined | 2
  Missing | 1

41. Secondary Outcome: Number of Participants With Polymorphisms in Aurora A Kinase
Time Frame: Cycle 1 Day 1 predose
Population: As per protocol amendment, no data was collected for polymorphisms in Aurora A Kinase.
Arm/Group | Alisertib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose (up to 422 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part 1 PIC Dose Escalation: Alisertib 25 or 35 mg, Powder-in-Capsule (PIC) formulation, orally, once daily (QD) for 21 days followed by a 7-day recovery period in 28-day cycles or alisertib 35, 45, 65 or 90 mg PIC, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 14 cycles). All participants received an initial starting dosage of alisertib PIC 25 mg, orally, twice daily (BID) on Day 1 (loading dose), followed by their respective dosage assignment.
- Part 1 ECT Dose Escalation: Alisertib 40 mg, Enteric-coated Tablet (ECT) formulation, orally, QD for 14 days followed by a 14-day recovery period in 28-day cycles, or alisertib 30, 40 or 50 mg ECT, orally BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 15 cycles).
- Part 2 PTCL: Participants with peripheral T-cell lymphoma (PTCL) received alisertib 50 mg ECT, orally, BID for 7 days followed by a 14-day recovery period in 21-day cycles, until disease progression or unacceptable alisertib-related toxicity (up to 2 cycles).
Arm/Group | Part 1 PIC Dose Escalation | Part 1 ECT Dose Escalation | Part 2 PTCL
Serious Adverse Events (participants affected / at risk) | 12/28 | 15/28 | 2/2
Other Adverse Events (participants affected / at risk) | 28/28 | 28/28 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 PIC Dose Escalation (N=28) | Part 1 ECT Dose Escalation (N=28) | Part 2 PTCL (N=2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — One treatment-emergent death occurred during treatment with alisertib 65 mg and was not related.
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — One treatment-emergent death occurred during treatment with alisertib 90 mg and was not related.
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — One treatment-emergent death occurred during treatment with alisertib 65 mg and was not related.
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) — One treatment-emergent death occurred during treatment with alisertib 50 mg and was not related.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 PIC Dose Escalation (N=28) | Part 1 ECT Dose Escalation (N=28) | Part 2 PTCL (N=2)
Neutropenia (Blood and lymphatic system disorders) | 13 (21) | 18 (35) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (14) | 13 (16) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 11 (15) | 12 (18) | 2 (5)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 11 (22) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 6 (9) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 14 (20) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (13) | 9 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 6 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 10 (11) | 10 (13) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1)
Chills (General disorders) | 4 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (8) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 5 (5) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 4 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Nutritional condition abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 6 (6) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (6) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (3) | 0 (0)
Eye disorders (Eye disorders) | 4 (5) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 2 (3) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.